CLINICAL TRIAL: NCT03416257
Title: Gut Microbial-related Choline Metabolite Trimethylamine-N-oxide is Associated With Progression of Carotid Artery Atherosclerosis in HIV Infection
Brief Title: TMAO and Atherosclerosis in HIV
Status: Completed | Type: Observational
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Qibin Qi, Assistant Professor, Albert Einstein College of Medicine
Other Study IDs: 2015-5145; K01HL129892 (NIH)
Record Dates: First submitted 2018-01-24; First posted 2018-01-31 (Actual); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Carotid Artery Plaque
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- WIHS: Women's Interagency HIV Study
  Interventions: Other: No intervention
- MACS: Multicenter AIDS Cohort Study
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
In the present study, the investigators sought to prospectively examine the associations of plasma levels of TMAO (trimethylamine oxide), choline, betaine, dimethylglycine, and sarcosine with risk of incident carotid artery plaque, assessed by repeated B-mode carotid artery ultrasound imaging over a 7-year period, in women and men with and without HIV infection from the WIHS (Women Interagency HIV Study) and MACS (Multicenter Aids Cohort Study).

ELIGIBILITY:
Inclusion Criteria:

* participants who underwent carotid artery imaging for plaque assessment at a baseline visit (2004-2006) and at a follow-up visit (2011-2013).

Exclusion Criteria:

* a history of coronary heart disease, individuals with prevalent diabetes or prevalent carotid artery plaques at baseline

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A total of 737 women and men with available baseline plasma choline metabolite data were included in this analysis. There were 520 HIV-infected (291 women, 229 men) and 217 HIV-uninfected (107 women, 110 men) participants included in this study. Baseline characteristics are shownin Table 1. HIV-infected and HIV-uninfected participants were generally similar in terms of demographic and behavioral variables, although HIV-infected participants were more likely to have a history of HCV infection. In addition, HIV-infected participants had lower total cholesterol and HDL cholesterol levels compared to those without HIV infection. The majority of HIV-infected individuals reported using potent ART at baseline (74% in women and 83% in men), and 46% of women and 66% of men had undetectable HIV-1 viral load (≤80 copies/mL). Compared to men, women were younger, more likely to be of black race or Hispanice thnicity and current smokers, and have a history of HCV infection and higher BMI.
Sampling Method: Non-Probability Sample
Enrollment: 737 (Actual)
Dates: Start 2004-04-12 (Actual); Primary Completion 2013-09-01 (Actual); Study Completion 2017-04-04 (Actual)

PRIMARY OUTCOMES:
incident carotid artery plaque | 2011-2013
  assessed by repeated B-mode carotid artery ultrasound imaging

IPD SHARING:
Plan to Share IPD: No